CLINICAL TRIAL: NCT03132818
Title: Impact of the Assumption in Charge of Medical Aid to the Procreation With Donation of Gametes on the Sexuality of the Couple
Acronym: SEXODON
Status: Withdrawn | Type: Observational
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-25 Dr Scheffler
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Sexuality
Keywords: Procreation with donation
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients undergoing AMP with oocyte donation
  Interventions: Other: To evaluate the prevalence of sexual disorders in patients receiving AMP
- Couples supported in AMP with sperm donation
  Interventions: Other: To evaluate the prevalence of sexual disorders in patients receiving AMP
- Couples supported in AMP intra torque
  Interventions: Other: To evaluate the prevalence of sexual disorders in patients receiving AMP

INTERVENTIONS:
Other: To evaluate the prevalence of sexual disorders in patients receiving AMP — To evaluate the prevalence of sexual disorders in patients receiving AMP

SUMMARY:
Sexual disorders associated with medical aid for procreation have already been demonstrated in several studies. However, few of them are interested in the problem of patients in charge of donating gametes, and if studied, it is often restricted to donating sperm to a small number of patients. For this reason, it would be interesting to study the impact of the intake and in charge and the treatments of the Medical Aid to the Procreation on this population of patients (including the patients treated in donation of sperm but also Those supported in oocyte donation)

ELIGIBILITY:
Inclusion Criteria:

* Couple, male and female, meeting the legal criteria for access to medically assisted procreation: a couple, a woman under the age of 43, who can testify to a life together. Then breakdown into 3 inclusion groups:

  * Group 1: Patients undergoing AMP with oocyte donation
  * Group 2: couples supported in AMP with sperm donation
  * Group 3: torque supported in intra torque AMP.

Exclusion Criteria:

* Patients who do not meet the legal criteria for access to the MPA.
* Patients in charge of Medical Assistance for Procreation "Viral Risk"
* Patients undergoing medical aid for procreation for pre-existing sexual dysfunction.
* Patients awaiting embryo reception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing AMP with donation of gametes whose objective is to detect and evaluate the prevalence of sexual disorders
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Analysis of anonymous sexual well-being questionnaires: one reserved for men, another reserved for women | 1 year
  Analysis of anonymous sexual well-being questionnaires: one reserved for men, another reserved for women

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France